CLINICAL TRIAL: NCT01397942
Title: Maximising the Taste and Health Value of Plant Food Products - Impact on Vegetable Consumption, Consumer Preferences and Human Health Factors.
Brief Title: Maximising the Taste and Health Value of Plant Food Products
Acronym: MAXVEG
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Aarhus University Hospital (Other)
Responsible Party: Principal Investigator, Per Bendix Jeppesen, Associate prof., PhD, Aarhus University Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 09-067129
Record Dates: First submitted 2011-07-18; First posted 2011-07-20 (Estimated); Last update posted 2015-03-11 (Estimated); Status verified 2015-03

CONDITIONS: Type 2 Diabetes
Keywords: Diet intervention; Type 2 diabetes; Vegetables; Phytochemicals
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Vegetables

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Diet intervention - Ancient vegatables (Experimental): A healthy Nordic diet with high content of bitter strong tasting vegetables and cabbages.
  Interventions: Other: Diet intervention
- Control Nordic diet (No Intervention): A diet habitually consumed in the Nordic countries
- Diet intervention - Modern Vegetables (Experimental): A healthy Nordic diet with high content of sweet and mild tasting vegetables and cabbages.
  Interventions: Other: Diet intervention

INTERVENTIONS:
Other: Diet intervention — The participants in the two experimental arms will each have to consume 500 g of vegetables and cabbages daily.
  Other Names: Vegetables; Ancient; Cabbages; Type 2 diabetes
  Arms: Diet intervention - Ancient vegatables; Diet intervention - Modern Vegetables

SUMMARY:
To investigate if a high dietary intake of bitter and strong tasting vegetables have positive health effects (insulin sensitivity, glucose tolerance, central obesity, fasting and postprandial lipid profile, blood pressure, vitamin D status and inflammatory markers, biomarkers of oxidative stress) on subjects with T2D. Also to look at a high dietary intake of mild and sweet modern vegetables or a normal western diet.

DETAILED DESCRIPTION:
The metabolic syndrome (MS), type 2 diabetes (T2D) and obesity are the world's most prevalent lifestyle diseases. This unfortunate development is mainly caused by lifestyle choices leading to obesity due to physical inactivity and excessive calorie intake.

Vegetables are an important part of the human diet and a major source of biologically active substances which determine the nutritional quality of food, color, taste, smell, antioxidative, anticarcinogenic, antihypertensive, anti-inflammatory, antihyperglycemia, immunostimulating and cholesterol-lowering properties.

Diet, as one aspect of lifestyle, is thought to be one of the modifiable variable risk factors for the development of MS and T2D, but more information is needed as to which components of the diet could be protective for the development and progression of MS and T2D with all its complications.

The study will be carried out as a 3-month randomized controlled parallel intervention study involving 60 subjects with T2D. During the fall year 2011 30 (10 in each group) subjects will participate and the remaining 30 subjects (10 in each group) in the fall 2012. The subjects will be randomized into 3 different diets:

1. A) "A healthy Nordic diet" with high content of bitter strong tasting vegetables and cabbages.
2. B) "A healthy Nordic diet" with high content of sweet and mild tasting vegetables and cabbages.
3. C) A diet habitually consumed in the Nordic countries (normal control diet). The subjects in groups A and B will each have to consume 500 g root vegetables and cabbages daily which will be handed out once a week. The participants will visit the study clinic at screening, and then once weekly during the intervention period (12 weeks). Beside the screening examination there will be 3 major visits (0, 6 and 12 weeks) where the participants will collect urine samples, complete a 3-day weighed food diary (to control diet intake) and undergo clinical examination incl. measuring of blood pressure, body composition and collection of fasting blood samples i.e. glucose, insulin, glucagon, HbA1c, GLP-1, lipids (triglycerides, HDL-, LDL- and total cholesterol), cytokines, adipokines, parathyroid hormone and vitamin D. During first (week 0) and third (week 12) major visit a 120 minutes oral glucose tolerance test is included collecting blood to analyze for glucose, insulin and triglycerides.

The study will contribute to the understanding on the impact of a diet with a high level of root vegetables and cabbages with either high or low levels of phytochemicals. Furthermore, the results can be used to develop new recommendations targeted T2D and MS subjects, and thereby contribute to a healthier lifestyle and to prevent any further development and progression of these lifestyle diseases. The overall perspective of the MAXVEG project is to enhance the consumption and production of bitter and strong tasting health promoting root vegetables and cabbages with high phytochemical content and high consumer preferences targeted specific consumer groups

ELIGIBILITY:
Inclusion Criteria:

* Type 2 diabetes in diet treatment or on oral anti-diabetic drug or the metabolic syndrome.

Exclusion Criteria:

* Other severe diseases or in treatment with insulin, GLP-1 analogs, glitazones.

Ages: 30 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 92 (Actual)
Dates: Start 2011-05; Primary Completion 2014-12 (Actual); Study Completion 2015-01 (Actual)

PRIMARY OUTCOMES:
Insulin sensitivity | 2 years
  Measured as the AUC from an Oral Glucose Tolerance Test

SECONDARY OUTCOMES:
Urine and blood samples | 2 years
  The fasting blood samples will be analyzed for: glucose, insulin, glucagon, HbA1c, lipids (triglycerides, HDL-, LDL- and total cholesterol), cytokines (, adipokines biomarkers of oxidative stress parathyroid hormone, vitamin D and GLP-1.
  Urine samples for metabolomics (isoprostanes and water-soluble metabolites).

CONTACTS AND LOCATIONS:
Overall Officials: Per B Jeppesen, Prof. PhD, Principal Investigator — University of Aarhus
Locations (1):
- Hospital Vendsyssel, Center for Clinical Research, Hjørring, North Denmark, Denmark

REFERENCES:
- See also: Click here for more information about this study: Maximising the Taste and Health Value of Plant Food Products (MAXVEG) — http://www.maxveg.dk